CLINICAL TRIAL: NCT07390877
Title: Cognitive and Metacognitive Remediation in Addiction Treatment: Randomized Controlled Trial of Efficacy in Parallel Arms
Acronym: R'COMET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC25_0044
Record Dates: First submitted 2025-12-05; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol use disorder; Cognitive remediation; Self-efficacity
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: This is a controlled study in which participants are randomized into two parallel groups: cognitive remediation group (R'COMET) or relaxation group (comparator).
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R'COMET treatment program (cognitive remediation program) (Experimental): The program will include 10 weekly sessions in an open group format to facilitate the patient's engagement in the treatment program (the patient may join the group at any time). The sessions will last 2 hours, ideally with 4-5 patients per session.
  Each session will include group and/or individual cognitive exercises to encourage interaction and the sharing of experiences, while also providing individualized and tailored support for each participant. Every cognitive exercise will be approached from a motivational perspective. The exercises offered during the sessions will be combined with systematic verbalization of strategies and emotional states, as well as psychoeducational, body-based, non-verbal communication, and cognitive-behavioral techniques. The proposed strategies will draw on both retrieval and compensatory approaches depending on the individual profiles.
  A progress booklet will be given to the patient.
  Interventions: Behavioral: cognitive remediation group
- Relaxation control program (Active Comparator): The relaxation program consists of 10 weekly sessions lasting 2 hours, held in open groups of 4 to 5 participants. Each session follows a flexible structure with several phases: a welcome moment where participants identify and express their feelings, a musical listening period to help them settle into the session, and a self-massage activity to promote bodily awareness. This is followed by a guided relaxation phase-either passive or active-to encourage physical and mental release. At the end of the session, a different breathing exercise is introduced each week so participants can discover which technique suits them best. The session concludes with a verbalization period, allowing everyone to share their sensations and impressions in a supportive, non-judgmental environment. Participants are encouraged to practice the exercises independently as well .
  Interventions: Behavioral: Relaxation control program

INTERVENTIONS:
Behavioral: cognitive remediation group — The program will include 10 weekly sessions in an open group format to facilitate the patient's engagement in the treatment program (the patient may join the group at any time). The sessions will last 2 hours, ideally with 4-5 patients per session.
  Each session will include group and/or individual cognitive exercises to encourage interaction and the sharing of experiences, while also providing individualized and tailored support for each participant. Every cognitive exercise will be approached from a motivational perspective. The exercises offered during the sessions will be combined with systematic verbalization of strategies and emotional states, as well as psychoeducational, body-based, non-verbal communication, and cognitive-behavioral techniques. The proposed strategies will draw on both retrieval and compensatory approaches depending on the individual profiles.
  Arms: R'COMET treatment program (cognitive remediation program)
Behavioral: Relaxation control program — The relaxation program consists of 10 weekly sessions lasting 2 hours, held in open groups of 4 to 5 participants. Each session follows a flexible structure with several phases: a welcome moment where participants identify and express their feelings, a musical listening period to help them settle into the session, and a self-massage activity to promote bodily awareness. This is followed by a guided relaxation phase-either passive or active-to encourage physical and mental release. At the end of the session, a different breathing exercise is introduced each week so participants can discover which technique suits them best. The session concludes with a verbalization period, allowing everyone to share their sensations and impressions in a supportive, non-judgmental environment. Participants are encouraged to practice the exercises independently as well .
  Arms: Relaxation control program

SUMMARY:
Cognitive and metacognitive remediation in addiction treatment: Value of Adding a cognitive remediation program to improve overall self-efficacy in patients with alcohol use disorder.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is the third leading risk factor for morbidity worldwide and represents a major public health issue. It is associated with numerous somatic and psychological harms, as well as cognitive impairments that lead to a deterioration in quality of life and continued AUD. It is therefore essential that cognitive disorders be targeted for treatment, along with craving, emotional dysregulation, and erroneous beliefs. Similarly, strengthening the sense of self-efficacy plays a crucial role in the recovery of patients with AUD and helps consolidate their ability to cope with the challenges of daily life. Several studies have demonstrated the benefits of cognitive remediation, and the need to offer this type of care more systematically has been widely advocated in several literature reviews. Based on data from the literature and validated cognitive remediation programs, the R'COMET program was designed for patients with SUD. It combines cognitive remediation, emotion perception, and metacognition. The aim of this program is to improve cognitive and metacognitive functions and to enhance the sense of self-efficacy, which is a major determinant of recovery in addictive disorders.

The objective of the R'COMET study is to evaluate the effectiveness of this program on overall self-efficacy, cognitive and metacognitive performance, alcohol consumption, and quality of life in patients with AUD, at the end of the program and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 (inclusive).
* Native French speaker or educated in French.
* Primary diagnosis of AUD according to DSM-5, with or without comorbid SUD.
* Currently in withdrawal: abstinent for at least 7 days and no more than 30 days.
* At least mild cognitive impairment, as measured by the BEARNI scale (mild impairment on the global scale or score below the threshold on at least one of the subtests).

Exclusion Criteria:

* Guardianship.
* Simultaneous participation in a cognitive rehabilitation group, an ETP programme or a mindfulness meditation group.
* Presence of unstabilised psychiatric or addictive comorbidity. The notion of instability is assessed over the past month and is defined by: (i) the need to introduce a new psychotropic treatment, (ii) the need to increase the dosage of an existing psychotropic treatment, (iii) the need for hospitalisation. Given the profile of the patients sought, the start of psychotropic treatment or hospitalisation to support alcohol withdrawal will not be considered exclusion criteria.
* Presence of neurodegenerative disease, Korsakoff's syndrome, mental retardation, or any other condition that may significantly interfere with the completion of assessments, as determined by the clinician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in General Self-Efficacy (SGSES-fr) | 6 months
  The primary outcome measure will be the change in the overall score on the SGSES-fr scale between the pre-treatment assessment (V1) and the immediate post-treatment assessment (V2). The advantage of this scale over other self-efficacy scales is that it is not linked to specific situations or behaviors, but represents a general measure.
  The minimum value is 10 and the maximum value is 40. 10 is a high outcome 40 is a low outcome It is expected that this score will increase between V1 and V2.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie TOUATI-HUREAU, Principal Investigator — Nantes University Hospital
Locations (6):
- France (6):
  - EPSM Epsylan, Blain
  - EPSM Georges Daumézon, Bouguenais
  - CHRU Brest, Brest
  - HIA, Brest
  - CHU de Nantes, Nantes
  - EPSM du Finistère Sud, Quimper

IPD SHARING:
Plan to Share IPD: No